CLINICAL TRIAL: NCT06170671
Title: Observational, Secondary Data Collection Study to Describe Acalabrutinib Treatment Outcomes in Chronic Lymphocytic Leukemia Patients in Real-life Setting in Romania
Brief Title: REAl-world Outcomes in CHronic Lymphocytic Leukemia Patients Receiving Acalabrutinib in Romania
Acronym: REACH
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8220R00055
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Cohort 1: December 2023 - collecting data retrospectively from patients routinely initiated on acalabrutinib between January - December 2023
  Interventions: Drug: Non interventional study
- Cohort 2: December 2024-collecting data retrospectively from patients routinely initated on acalabrutinib between January - December 2024
  Interventions: Drug: Non interventional study

INTERVENTIONS:
Drug: Non interventional study — CLL patients routinely initiated on acalabrutinib by their physician between January 2023 -December 2024. Retrospective secondary data collection

SUMMARY:
Acalabrutinib received European Medicines Agency approval on November 2020 for for CLL adult patients, either as monotherapy or in combination with obinutuzumab, in previously untreated patients or as monotherapy in patients who have received at least one prior therapy and is reimbursed in Romania since January 2023. In the absence of disease registries or national datasets patient population receiving acalabrutinib in real life setting is not well characterized. The study aims to look into this population outcomes and clinical characteristics having as primary objective time to discontinuation by line of treatment and secondary objectives: reasons for discontinuation, effectiveness of acalabrutinib in real-life practice, baseline clinical and demographic characteristics, treatment patterns and major determinants of treatment discontinuation. The study will retrospectively collect longitudinal data from 250 patients at national level,at pre-defined timepoints for 3 years, from 2 sequential cohorts,1st one enrolled on December 2023 and 2nd one enrolled in December 2024 based on the acalabrutinib start year..

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age >18 years) with confirmed diagnosis of chronic lymphocytic leukemia/ small lymphocytic lymphoma
* Patients initiating front-line or subsequent treatment with acalabrutinib between January 2023 and Dec 2024 according to the national therapeutic protocol
* Patients able and willing to provide their written informed consent to participate in the study

Exclusion Criteria:

* The treatment with acalabrutinib was initiated during an interventional clinical trial
* Enrolment performed less than 30 days from start of treatment with acalabrutinib

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CLL patients routinely initiated on acalabrutinib in front-line or subsequent treatment during the study eligibility window January 2023-December 2024
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Time to acalabrutinib treatment discontinuation (TTD) | Once a year during the 3 years of follow up since acalabrutinib start
  TTD is defined as the time between the first day of acalabrutinib treatment and the day that acalabrutinib is definitely stopped for whatever reason or death

SECONDARY OUTCOMES:
Reasons for treatment discontinuation | Once a year until end of the study ( 3 years from start of acalabrutinib)
  Reasons for acalabrutinib interruption
effectiveness of acalabrutinib | Once a year until end of the study ( 3 years from start of acalabrutinib)
  Real world progression free survival (rwPFS) is defined as the time from initiation of acalabrutinib therapy (index date) until earliest record of disease progression determined by physicians' assessment (clinical or radiological progression or start of a new line therapy),or death
Baseline clinical and demographic characteristics | At first data collection for cohort 1 in December 2023 and at first data collection for cohort 2 in December 2024
  Demographic characteristics (age,gender, BMI) and disease characteristics (age at diagnosis, staging, symptoms, active disease criteria,previous treatment
acalabrutinib interruption | Once a year until end of the study (3 years from the start of acalabrutinib)
  Percentage of patients with acalabrutinib interruption
time to interruption | Once a year until end of the study ( 3 years from start of acalabrutinib)
  Time between first day of acalabrutinib and the day of first interruption of acalabrutinib
duration of interruption | once a year until the end of the study ( 3 years from acalabrutinib start)
  Time between the first day of acalabrutinib interruption and the first day of acalabrutinib restart
acalabrutinib dose changes | once a year until the end of the study ( 3 years from acalabrutinib start)
  Percentage of patients with dose changes
Reasons of acalabrutinib dose changes | once a year until the end of the study ( 3 years from acalabrutinib start)
  Reasons of acalabrutinib dose changes (all including adverse events)
Major determinant of treatment discontinuation | once a year until end of the study( 3 years from acalabrutinib start)
  a multivariate analysis (Cox model) will be performed to study correlation between TTD and patient characteristics at baseline.

CONTACTS AND LOCATIONS:
Locations (14):
- Romania (14):
  - Research Site, Piteşti, Argeş
  - Research Site, Oradea, Bihor County
  - Research Site, Cluj-Napoca, Cluj
  - Research Site, Craiova, Dolj
  - Research Site, Deva, Hunedoara County
  - Research Site, Baia Mare, Maramureş
  - Research Site, Târgu Mureş, Mureș County
  - Research Site, Piatra Neamţ, Neamț County
  - Research Site, Timișoara, Timiș County
  - Research Site, Focşani, Vrancea
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Galati
  - Research Site, Iași

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
  Supporting
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home